CLINICAL TRIAL: NCT00290823
Title: Treatment of Intraparenchymal Neurocysticercosis: Effect of Increased Dosing of Corticosteroids on Seizure Frequency
Brief Title: Corticosteroids to Reduce Frequency of Seizures in Neurocysticercosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05IN214; 05-I-N214; NCT00344396 (obsolete NCT alias)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Neurocysticercosis
Keywords: Taenia; Seizures; Tapeworm; Parasite
MeSH Terms: conditions — Neurocysticercosis; Seizures; Cestode Infections | interventions — Albendazole; Dexamethasone; Omeprazole

ARMS (2):
- 1 (Experimental): Participants will receive 6 mg dexamethasone daily for 10 days Participants will also receive albendazole and omeprazole.
  Interventions: Drug: Albendazole; Drug: Dexamethasone; Drug: Omeprazole
- 2 (Experimental): Participants will receive 6 mg dexamethasone daily for 10 days, then 8 mg dexamethasone daily for 4 weeks with a 2-week taper. Participants will also receive albendazole and omeprazole.
  Interventions: Drug: Albendazole; Drug: Dexamethasone; Drug: Omeprazole

INTERVENTIONS:
Drug: Albendazole — 400 mg tablet taken orally twice daily
Drug: Dexamethasone — 6mg or 8mg taken daily
Drug: Omeprazole — 20 mg tablet taken orally daily

SUMMARY:
The purpose of this study is to determine whether a short course of increased corticosteroid dosing with tapered dosing decreases seizure frequency as compared to standard corticosteroid dosing in patients with neurocysticercosis (NCC).

DETAILED DESCRIPTION:
NCC is the most common parasitic infection of the central nervous system (CNS). It is caused by ingestion of eggs from a tapeworm of genus Taenia. Inflammation, seizures, or neurologic problems may occur in a patient with NCC. Corticosteroids are the current standard of care for NCC patients, but corticosteroids have many side effects. Albendazole is used to treat infections caused by worms; however, it is unclear if its use with the corticosteroid dexamethasone will decrease seizure frequency in NCC patients. The purpose of this study is to evaluate the efficacy of reducing seizure frequency with a short course of dexamethasone with tapered dosing when given with albendazole, as compared to standard dexamethasone and albendazole treatment, in NCC patients.

In this open label study, patients will be randomly assigned to one of two arms. Group I will receive 6 mg dexamethasone daily for 10 days only. Group II will receive 6 mg dexamethasone daily for 10 days, then 8 mg dexamethasone daily for 4 weeks with a 2-week taper. Both groups will also receive albendazole and omeprazole (a medicine that helps prevent gastroesophageal disease [GERD], a side effect of corticosteroid use). There will be 13 study visits over a 360-day period. Blood collection will occur at most visits. Group II will also undergo sputum smears and rapid culture testing on Days 14, 28, and 42. Patients will undergo magnetic resonance imaging (MRI) at screening and on Day 180 and computed tomography (CT) scanning on Day 360.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with intraparenchymal NCC with 20 or fewer active cysts, as confirmed by enzyme-linked immunoelectrotransfer blot (EITB)
* Diagnosed with epilepsy secondary to NCC, with history of one or more spontaneous seizures within the 6 months prior to study entry
* Willingness to be hospitalized for a minimum of 2 weeks for this study
* PPD negative OR negative smears for tuberculosis (TB) if PPD positive
* Willing to use acceptable forms of contraception during the study and for at least 1 month after albendazole therapy

Exclusion Criteria:

* Primary generalized seizures not caused by NCC
* Subarachnoid or ventricular NCC
* Any vesicular lesion greater than 2 cm in diameter
* Previous therapy with albendazole or praziquantel within 2 years of study entry. Patients who have previously received single-dose albendazole for intestinal parasites are not excluded.
* Intracranial hypertension, as confirmed by CT or MRI
* History of status epilepticus
* Focal neurological defects
* Unstable or consistently abnormal vital signs (e.g., body temperature, pulse, respiratory rate, blood pressure)
* Cysts in critical regions, including brainstem or the eyes
* Pulmonary TB
* History of TB in the patient or history of TB in close contact of patient
* Chest x-ray suggestive of past or current TB
* Diabetes
* Systemic conditions (e.g., chronic kidney failure, liver disease, heart failure, steroid-dependent immune diseases) other than NCC that may interfere with the study
* Predicted survival time of less than 1 year
* Inability to undergo CT or MRI
* Hypersensitivity to albendazole, antiepileptic drugs, or contrast
* Hypertension at rest
* Require corticosteroids, received corticosteroids in the 4 weeks prior to study entry, or received corticosteroids for 9 or more days within the 6 months prior to study entry
* Other CNS processes that may interfere with study assessments
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2006-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cumulative frequency of partial, generalized, and total seizures | Through Day 42

SECONDARY OUTCOMES:
Cumulative frequency of generalized seizures | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Theodore E. Nash, MD, Principal Investigator — Gastrointestinal Parasites Section, Laboratory of Parasitic Diseases, NIAID; Hector H. Garcia, MD, PhD, Study Director — Department of Microbiology, Universidad Peruana Cayetano Heredia
Locations (1):
- Instituto Especializado en Ciencias Neurologicas, Lima, Peru

REFERENCES:
- [Background] Del Brutto OH. Neurocysticercosis. Semin Neurol. 2005 Sep;25(3):243-51. doi: 10.1055/s-2005-917661. PMID 16170737
- [Background] Garcia HH, Gilman R, Martinez M, Tsang VC, Pilcher JB, Herrera G, Diaz F, Alvarado M, Miranda E. Cysticercosis as a major cause of epilepsy in Peru. The Cysticercosis Working Group in Peru (CWG). Lancet. 1993 Jan 23;341(8839):197-200. doi: 10.1016/0140-6736(93)90064-n. PMID 8093496
- [Background] Medina MT, Rosas E, Rubio-Donnadieu F, Sotelo J. Neurocysticercosis as the main cause of late-onset epilepsy in Mexico. Arch Intern Med. 1990 Feb;150(2):325-7. PMID 2302008